CLINICAL TRIAL: NCT01597609
Title: A Single-blind, Randomised, Placebo-controlled, Parallel Group, Incomplete Block Design, Benchmark Study to Characterise the Physiology of Weight Loss and Regain Under Dietary, Behavioural and Pharmacological Interventions in Healthy Obese Subjects
Brief Title: A Study to Characterise the Physiology of Weight Loss and Regain Under Dietary, Behavioural and Pharmacological Interventions in Healthy Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 110739
Record Dates: First submitted 2012-04-12; First posted 2012-05-14 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — sibutramine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A (Experimental): - 600 Kcal deficit, Sibutramine placebo
  Interventions: Other: sibutramine placebo
- Cohort B (Experimental): - 600 Kcal deficit, Sibutramine 10 mg once daily
  Interventions: Drug: sibutramine
- Cohort C (Experimental): - 600 Kcal deficit, Moderate exercise (The energy expenditure will be equivalent to 30 minutes of brisk walking/5 times week i.e. ~1,000 Kcal/week) /sibutramine placebo
  Interventions: Other: sibutramine placebo

INTERVENTIONS:
Drug: sibutramine — 10 mg, taken orally once per day for 12 weeks
  Arms: Cohort B
Other: sibutramine placebo — taken orally once per day for 12 weeks
  Arms: Cohort A; Cohort C

SUMMARY:
Approximately 60 obese, but otherwise healthy, subjects will be assessed in this benchmark study to investigate the physiological changes associated with weight loss and regain. The aim is to estimate the changes in body composition during and after three interventions (i) calorie restricted diet + a marketed anti-obesity drug (sibutramine )(ii) calorie restricted diet + sibutramine placebo, and (iii) calorie restricted diet + moderate exercise. The interventions will last 12 weeks, after which there is a further 12 week observation period during which subjects will return to their normal lifestyle and are expected to regain weight. Additionally, a range of biomarkers may be evaluated to determine whether there are correlations at early and late time points with weight and fat loss and weight and fat regain. The changes in body composition and other biomarkers will be used to determine whether mathematical models can be built that predict the weight loss and regain of individual subjects. In addition, the usefulness of tools that may aid the physiological characterisation of weight loss/regain will be assessed, in particular methods for measuring energy expenditure and energy intake such as ambulatory activity meter, Sussex Ingestion Pattern Monitor ™ (SIPM), hunger-satiety VAS, indirect calorimetry and, if available, the Theranos in-home graphical user interface (GUI) portal. Knowledge of the body composition changes resulting from these typical weight loss interventions and predictive markers of response would facilitate the design of future studies for novel anti-obesity agents and allow earlier, more informed triaging of NCEs.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy male or female adult subject aged 20 to 55 years, inclusive.

Subjects will be allowed in the study if they have medical conditions, such as asthma, which will not compromise the validity of the study in the opinion of the Principal Investigator and Medical Advisor.

* BMI within the range 30.0 to 40.0 kg/m2 inclusive.
* Has been obese from approximately the age of 18 or above.
* Has demonstrated previous weight loss sustained for a minimum of one month.
* Pre-menopausal female subjects of child bearing potential who are not pregnant or breast feeding will be eligible to participate if they comply with the following: Abstinence.

The lifestyle of female subjects should be such that there is complete abstinence from intercourse from at least 30 days prior to receiving study medication and to continue until 30 days beyond the last study event, or 5 half lives of the study medication, whichever is the longest. If a subject claims abstinence as their method of contraception, they must agree to use a double barrier method (condoms, cervical/vault cap or diaphragm plus spermicide) should they become sexually active during the time frame described above. One of the following methods is acceptable as the sole method of contraception if there is indisputable data that it is >99% effective, otherwise it should be used with a barrier method (condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicidal foam/gel/film/cream/suppository): Documented tubal ligation, IUD or IUS, Oral contraception, Male partner sterilization (vasectomy) at least 6 months prior to the female subject's entry into the study and is the sole partner for that female subject. Condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository (Appendix 3).

* Subject has provided signed and dated, written informed consent prior to enrolment in the study.
* The subject is able to understand and comply with protocol requirements, instructions, and protocol-stated restrictions.

Exclusion Criteria:

* Has either a previous disease or current medical condition, which as judged by the Investigator, may affect the interpretation of data. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease or endocrine disease.
* Currently has closed angle glaucoma.
* Has prostatic hypertrophy or hyperplasia.
* Females who are post-menopausal (post-menopausal females defined as being amenorrhoeic for more than 2 years with an appropriate clinical profile, e.g. history of vasomotor symptoms and confirmed by an FSH ≥ 40 mIU/mL).
* Known history of panic attacks and/or claustrophobia or other conditions precluding safe DEXA and Echo MRI-AH scans according to local guidelines, (e.g., pacemaker, hearing aid, metallic body piercing and/or other metal implants) or in the opinion of the Investigator the subject exceeds size limitations for the instruments.
* Has a history of clinically significant eating disorders (diagnosed and/or treated) such as previous anorexia nervosa, binge-eating disorder or bulimia nervosa.
* Has a recent history of weight loss (or gain) defined as a change of ≥ 5 % in the 3 months prior to screening.
* Has a history of being obese in childhood.
* Has had bariatric surgical intervention for obesity.
* Has a confirmed diagnosis of polycystic ovary syndrome.
* Has a history of alcohol or substance abuse or dependence in the 6 months prior to screening as determined by the Investigator. Abuse of alcohol, defined for males, as an average weekly intake of greater than 21 units (or an average daily intake of greater than 3 units), or defined for females, as an average weekly intake of greater than 14 units (or an average daily intake of greater than 2 units). One unit is equivalent to a half-pint (220mL) of beer or 1 (25mL) measure of spirits or 1 glass (125mL) of wine.
* Subjects will not be eligible if they plan to alter their current smoking (or other tobacco use) status during the course of the study, or if they have quit smoking less than 3 months prior to screening. Because of the effects of tobacco smoke on biomarkers, subjects may be classified as 'never smokers' or 'current smokers (abstaining at study visit) + former smokers'.
* Subjects who could not refrain from smoking during the time of the visit in the unit.
* Has a positive urine drug test at screening or pre-intervention. At a minimum, subjects will be screened for amphetamines, barbiturates, cocaine, opiates, cannabinoids, and benzodiazepines, and may be screened randomly throughout the study.
* Positive results for hepatitis C antibodies, hepatitis B surface antigen, or HIV at screening. If negative results have been obtained in the last 6 months, it is not necessary to repeat the tests unless indicated by clinical judgment.
* Has a documented history of hepatobiliary disease or hepatic enzyme elevation including any one of the following: ALT or AST > 2.5 times the upper limit of normal at screening or pre-intervention Total bilirubin > 1.5 times the upper limit of normal at screening or pre-intervention.

Subjects above this limit may only be included if direct bilirubin is within normal limits, which would be consistent with Gilbert's disease.

* Fasting triglycerides > 600mg/dL at screening or pre-intervention. If receiving lipidlowering therapy, then the subject must have been on stable doses for at least 3 months prior to screening.
* Has known type 1 or type 2 diabetes mellitus; or has fasting plasma glucose ≥ 126mg/dL (7.0 mmol/L) at screening. Subjects who fall outside this range but below 140 mg/dL fasting will be evaluated for inclusion by the PI or designee.
* Has a thyroid disorder that is not under adequate control with a stable dose of hormone replacement for at least 3 months prior to screening. Inadequate control is defined as a TSH level below the lower limit of the reference range (LLRR) or > 1.5

  × ULRR at screening.
* Has a systolic BP above 150 mmHg and/or diastolic BP above 90 mmHg at screening. If receiving anti-hypertensive therapy, then the subject must have been on stable doses for at least 3 months prior to screening.
* Is incapable or unwilling to participate in a moderate walking exercise program.
* Is pregnant or planning a pregnancy in the following 27 weeks from screening.
* Has any clinically significant abnormality identified on the medical or laboratory evaluation, including 12-lead ECG. A subject with a clinically significant abnormality or laboratory parameters outside the reference range for this age group may be included only if the Investigator considers that the finding will not introduce additional risk factors and will not interfere with the study procedures. Any questions regarding the significance of abnormal clinical findings in screening results should be discussed with the GSK Medical Monitor.
* Exclusions relating to concomitant preparations and medications: use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (which ever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and Sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Planning to commence or stop HRT or oral contraceptives during the course of the study. Female subjects who are taking an oral contraceptive preparation at the time of screening may be eligible for enrollment in the study.
* Use of weight loss drugs within 3 months of date of randomization.
* Use of any oral anti-diabetic medication. (including metformin, sulphonylureas, thiazolidinediones, GLP-1 agonist, DDPIV inhibitors).
* Use of anti-depressants (SSRI, tricyclic, bupropion etc) within 3 months of screening.
* Use of diuretics (other than stable dosing of HCTZ), systemic corticosteroids (inhaled and intranasal corticosteroids are permitted), or any other medication within 3 weeks prior to any scheduled dose of study medication that may result in electrolyte depletion.
* Use of warfarin, digoxin, oral anti-coagulants (other than aspirin and non-steroidal anti-inflammatory drugs), or antiretroviral medications.
* Use of macrolide antibiotics during the interventional part of the study.
* Use of any investigational drug or device during the study or in the 30 days prior to first dosing with study medication.
* History or presence of allergy or hypersensitivity to sibutramine or any of its components, or drugs of this class, or a history of drug or other allergy that, in the opinion of the primary investigator, contraindicates study participation.
* Has donated 500 or more milliliters of blood within 56 days prior to dosing or has the intention of donating blood the month after completing the study.
* Is unwilling to adhere to protocol-stated restrictions while participating in the study.
* The Investigator considers the subject unfit for the study as a result of the medical interview, physical examination, or screening investigations.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05-22 (Actual); Primary Completion 2010-03-04 (Actual); Study Completion 2010-03-04 (Actual)

PRIMARY OUTCOMES:
Measures of body composition (fat mass, lean mass and total body water) using Echo MRI-AH and DEXA during the intervention and follow-up phases | 24 Weeks
  estimate the changes during and after three interventions: (i) calorie restricted diet + a marketed anti-obesity drug (sibutramine), (ii) calorie restricted diet + sibutramine placebo, and (iii) calorie restricted diet + moderate exercise + sibutramine placebo
Measures of body weight and body mass index (BMI) during the intervention and follow-up phases. | 24 weeks
  estimate the changes during and after three interventions: (i) calorie restricted diet + a marketed anti-obesity drug (sibutramine), (ii) calorie restricted diet + sibutramine placebo, and (iii) calorie restricted diet + moderate exercise + sibutramine placebo
Measures of waist and hip circumference during the intervention and follow-up phases. | 24 weeks
  estimate the changes during and after three interventions: (i) calorie restricted diet + a marketed anti-obesity drug (sibutramine), (ii) calorie restricted diet + sibutramine placebo, and (iii) calorie restricted diet + moderate exercise + sibutramine placebo

SECONDARY OUTCOMES:
Mathematical models that use biomarkers of (i) body composition and metabolic status, (ii) macronutrient intake, and (iii) energy expenditure to predict later changes in weight and body composition during the intervention and follow-up phases. | 24 Weeks
  This will involve looking at the levels of a range of biomarkers including leptin and adiponectin.
Measures of energy expenditure | 24 Weeks
  using (i) an ambulatory activity meter, the ambulatory activity meter Armband, (ii) by indirect calorimetry using a ventilated hood, (iii) by self-reported diary entry and (iv) the Theranos GUI, if available, during the intervention and follow-up phases.
Measures of food intake, satiety and satiation | 24 Weeks
  using (i) food diaries, (ii) the Sussex Ingestion Pattern Monitor ™ (SIPM)), (iii) the Hunger, Craving, and Fullness Questionnaire (HCFQ/VAS), (iv) the Hunger/Satiety visual analogue scale and (iv) the Theranos GUI, if available, during the intervention and follow-up phases.
Measures of insulin sensitivity | 24 Weeks
  calculated from fasting insulin, glucose, free fatty acids and glycerol levels during the intervention and follow-up phases.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- See also: Results for study 110739 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/110739?search=study&search_terms=110739#rs